CLINICAL TRIAL: NCT03520426
Title: A Randomized Controlled Trial for the Evaluation of Efficacy and Safety of Votiva for Vaginal Rejuvenation
Brief Title: Evaluation of Efficacy and Safety of Votiva for Vaginal Rejuvenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walden, Jennifer L., M.D.,P.L.L.C. (Individual)
Collaborators: Aviva Preminger, MD., P.L.L.C. (Unknown); InMode MD Ltd. (Industry)
Responsible Party: Principal Investigator, Jennifer Walden, Jennifer L. Walden, MD, FACS, Walden, Jennifer L., M.D.,P.L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6198
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-04

CONDITIONS: Vaginal Atrophy; Vaginal Relaxation; Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Votiva RF (Experimental): Patients will undergo radiofrequency treatment using the Votiva FormaV and FractoraV hand pieces, using the device's standard protocol. Patients will have 3 treatments spaced 3-4 weeks apart and two follow-up visits. Duration of each treatment visit is approximately 1-1.5 hours. Prior to treatment and follow-up visit, each patient will be assessed using standardized photos, perineometry, and validated questionnaires.
  Interventions: Device: Votiva RF
- Votiva RF Sham (Sham Comparator): Patients will undergo the acts of receiving radiofrequency treatment with the Votiva FormaV and FractoraV hand pieces, but no direct energy will be applied. Patients will have 3 treatments spaced 3-4 weeks apart and 2 follow-up visits. Duration of each treatment visit is approximately 1-1.5 hours. Prior to treatment and follow-up visit, each patient will be assessed using standardized photos, perineometry, and validated questionnaires.
  Interventions: Device: Votiva RF

INTERVENTIONS:
Device: Votiva RF — The Votiva system is approved by the U.S. Food and Drug Administration for treatment of sexual dysfunction as well as in combination with Kegel exercises for tightening of the muscles of the pelvic floor to increase muscle tone. One part of the system, the fractora handpiece, is approved for tissue coagulation for the purpose of skin rejuvenation. The Votiva has two hand pieces, Forma and Fractora, which have been cleared by the United States Food and Drug Administration (FDA) and are used during dermatological procedures.

SUMMARY:
This is a multi-site, randomized, prospective study designed to evaluate the safety and efficacy of the Votiva device headpieces through radiofrequency for vaginal rejuvenation. An anticipated 50 subjects will undergo 3 treatments of the vulvovaginal area using radiofrequency unit or radiofrequency placebo. Study duration for each subject is approximately six months (including screening, 3 treatment sessions 3-4 weeks apart and 2 follow-up visit at 3 and 6 months post initiation of treatment (4 and 12 weeks after completion of last treatment). Efficacy will be measured and evaluated by validated questionnaires to include: The Vulvovaginal Symptoms Questionnaire, Vaginal Laxity Questionnaire (VLQ), Urogenital Distress Short Form (UDI-6) and Incontinence Impact Questionnaire Short Form (IIQ-7), Female Sexual Function Index (FSFI) and the Female Sexual Distress Scale-Revised (FSDS-R).

DETAILED DESCRIPTION:
Vaginal rejuvenation is a catch-all term of aesthetic and functional procedures which claim to provide relief of many issues affecting women's health, ranging from postmenopausal vulvovaginal symptoms (i.e. dryness, burning, itching), stress urinary incontinence, sexual dysfunction or discomfort, vaginal laxity, and external labial appearance, amongst others.1,2 Several companies have emerged with non-invasive or minimally-invasive technologies to alleviate these conditions which operate by radiofrequency (RF) delivery, Hybrid Fractional Laser, fractional CO2 laser3, or Er:YAG4. Votiva by InMode is unique in its usage as both an internal and external rejuvenating device.

The RF technologies work theoretically by heating the connective tissue of the vaginal wall to 40 to 42°C thereby remodeling extracellular matrix configuration. Once optimal temperatures are reached, collagen contraction, neocollagenesis, vascularization, and growth factor infiltration could lead to durable vaginal wall changes with improvement in elasticity and moisture of the vaginal wall. Although numerous studies have demonstrated the therapeutic efficacy of energy-based devices in rejuvenation of the face, neck, and décolleté, their application in the vaginal canal is a fairly new concept that is currently being studied.11

Given the paucity of data, this study aims to assess the utility and safety of the RF device Votiva in a two arm prospective case control trial for improvement in external labial appearance, vaginal laxity, sexual function and urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25-65 years with symptoms of vaginal relaxation syndrome and/or urinary incontinence who desire vaginal rejuvenation treatment.
* Informed Consent Form, Photo Release and sharing of assessments signed by the subject.
* Ability and willingness to follow the study visits schedule.
* Ability and willingness to adhere to prescribed medication regime.

Exclusion Criteria:

* Unable to commit to future appointments within one year
* Planning on moving away from the New York or Austin area within one year
* History of other energy-based vaginal therapy within one year
* Intermittent vaginal hormone replacement therapy. If patients are on hormone replacement therapy, they should maintain their dosing throughout the study. (If using systemic HRT, shouldn't change it during the whole study period)
* Prior labiaplasty
* Prior anti-incontinence surgery in the last 12 months
* Urinary incontinence requiring more than 2 pads/day
* Urinary tract infection in the past 3 months
* Immunodeficiency status (steroid intake, ongoing chemotherapy)
* Diffuse pain syndrome or chronic pain requiring daily narcotics
* Chronic vaginitis including bacterial vaginosis, HPV, herpes, or other active STI
* Abnormal Papanicolaou test result in the last 2 years
* Abnormal pelvic exam (i.e. concerning lesions) or anterior or posterior vaginal prolapse in the last 2 years
* Undiagnosed abnormal genital bleeding
* If of child-bearing potential or less than two years postmenopausal, not using a medically approved method of contraception (i.e. oral, transdermal, implanted contraceptives, intrauterine device, diaphragm, condom, etc.)
* If patients are using a Nuvaring, they must use an alternate form of contraception during the three treatment months
* Pregnancy (determined by urine HCG prior to procedure) or lactating
* Psychiatric conditions
* Pacemaker or internal defibrillator, or other implanted metallic or electronic device.
* Permanent implant in the treated area such as metal plates and screws or silicone.
* Current or history of any type of cancer, or pre-malignant conditions.
* Severe concurrent conditions, such as cardiac disorders.
* History of or current diseases stimulated by heat, such as recurrent Herpes Simplex, in the area of the vagina where the study device will be applied. This area may be included in the study only following a prophylactic regimen.
* Poorly controlled endocrine disorders, such as diabetes.
* Any active skin condition in the treatment area, such as sores, infection, eczema, and rash. History of skin disorders, keloids (irregularly shaped scars), abnormal wound healing, as well as very dry and fragile skin.
* History of a bleeding disorder in which the blood's ability to form clots is impaired.
* Any treatment or surgery performed in the treatment area within a year prior to treatment.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* Any therapies or medications which may interfere with the use of the study device.
* Compromised health as determined by the study doctor.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Sexual-impact of vulvovaginal symptoms in postmenopausal women | 6 months
  Assessed and measured by: The Vulvovaginal Symptoms Questionnaire (VVSQ)
Improved Vaginal Laxity | 6 months
  Vaginal laxity/tightness assessed and measured by: Vaginal Laxity Questionnaire (VLQ)
Improved Sexual Function | 6 months
  Sexual dysfunction assessed and measured by: Female Sexual Function Index (FSFI)
Measuring Sexually Related Personal Distress in Women With Female Sexual Dysfunction | 6 months
  Assess distress associated with impaired sexual function assessed and measured by: Female Sexual Distress Scale-Revised Questionnaire
Urogenital Distress Inventory | 6 months
  Assessed and measured by: Urogenital Distress Inventory, Short Form (UDI-6) scores
Urinary Incontinence Impact | 6 months
  Assessed and measured by: Incontinence Impact Questionnaire Short Form (IIQ-7)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L. Walden, MD, Principal Investigator — Owner; Aviva Preminger, MD, Principal Investigator — Co-Site PI
Locations (2):
- United States (2):
  - Preminger Plastic Surgery, New York, New York
  - Jennifer L. Walden MD., P.L.L.C., Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Millheiser LS, Pauls RN, Herbst SJ, Chen BH. Radiofrequency treatment of vaginal laxity after vaginal delivery: nonsurgical vaginal tightening. J Sex Med. 2010 Sep;7(9):3088-95. doi: 10.1111/j.1743-6109.2010.01910.x. PMID 20584127
- [Background] Sekiguchi Y, Utsugisawa Y, Azekosi Y, Kinjo M, Song M, Kubota Y, Kingsberg SA, Krychman ML. Laxity of the vaginal introitus after childbirth: nonsurgical outpatient procedure for vaginal tissue restoration and improved sexual satisfaction using low-energy radiofrequency thermal therapy. J Womens Health (Larchmt). 2013 Sep;22(9):775-81. doi: 10.1089/jwh.2012.4123. Epub 2013 Aug 16. PMID 23952177
- [Background] Zerbinati N, Serati M, Origoni M, Candiani M, Iannitti T, Salvatore S, Marotta F, Calligaro A. Microscopic and ultrastructural modifications of postmenopausal atrophic vaginal mucosa after fractional carbon dioxide laser treatment. Lasers Med Sci. 2015 Jan;30(1):429-36. doi: 10.1007/s10103-014-1677-2. Epub 2014 Nov 20. PMID 25410301
- [Background] Lee MS. Treatment of Vaginal Relaxation Syndrome with an Erbium:YAG Laser Using 90 degrees and 360 degrees Scanning Scopes: A Pilot Study & Short-term Results. Laser Ther. 2014 Jul 1;23(2):129-38. doi: 10.5978/islsm.14-OR-11. PMID 25071312
- [Background] Committee on Gynecologic Practice, American College of Obstetricians and Gynecologists. ACOG Committee Opinion No. 378: Vaginal "rejuvenation" and cosmetic vaginal procedures. Obstet Gynecol. 2007 Sep;110(3):737-8. doi: 10.1097/01.AOG.0000263927.82639.9b. PMID 17766626
- [Background] Alinsod RM. Transcutaneous temperature controlled radiofrequency for orgasmic dysfunction. Lasers Surg Med. 2016 Sep;48(7):641-5. doi: 10.1002/lsm.22537. Epub 2016 May 19. PMID 27197701
- [Background] Coad JE, Vos JA, Curtis A, Krychman M. Safety and mechanisms of action supporting nonablative radiofrequency thermal therapy for vaginal introitus laxity occurring in women after childbirth: Histological study in the sheep vaginal model. J Sex Med 2013;10(Supplement 2):175.
- [Background] Krychman M, Rowan CG, Allan BB, DeRogatis L, Durbin S, Yacoubian A, Wilkerson D. Effect of Single-Treatment, Surface-Cooled Radiofrequency Therapy on Vaginal Laxity and Female Sexual Function: The VIVEVE I Randomized Controlled Trial. J Sex Med. 2017 Feb;14(2):215-225. doi: 10.1016/j.jsxm.2016.11.322. PMID 28161079
- [Background] Karcher C, Sadick N. Vaginal rejuvenation using energy-based devices. Int J Womens Dermatol. 2016 Jun 21;2(3):85-88. doi: 10.1016/j.ijwd.2016.05.003. eCollection 2016 Sep. PMID 28492016
- [Background] Erekson EA, Yip SO, Wedderburn TS, Martin DK, Li FY, Choi JN, Kenton KS, Fried TR. The Vulvovaginal Symptoms Questionnaire: a questionnaire for measuring vulvovaginal symptoms in postmenopausal women. Menopause. 2013 Sep;20(9):973-9. doi: 10.1097/GME.0b013e318282600b. PMID 23481118
- [Background] Erekson EA, Li FY, Martin DK, Fried TR. Vulvovaginal symptoms prevalence in postmenopausal women and relationship to other menopausal symptoms and pelvic floor disorders. Menopause. 2016 Apr;23(4):368-75. doi: 10.1097/GME.0000000000000549. PMID 26645820
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Derogatis L, Clayton A, Lewis-D'Agostino D, Wunderlich G, Fu Y. Validation of the female sexual distress scale-revised for assessing distress in women with hypoactive sexual desire disorder. J Sex Med. 2008 Feb;5(2):357-64. doi: 10.1111/j.1743-6109.2007.00672.x. Epub 2007 Nov 27. PMID 18042215